CLINICAL TRIAL: NCT04935593
Title: Strengthening Social, Emotional and Behavioral Resilience: The RENEW (Resilience in Emotional and Behavioral Wellbeing) Pilot Randomized Controlled Trial
Brief Title: Strengthening Social, Emotional and Behavioral Resilience
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Taipei Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: pbowrin001
Record Dates: First submitted 2021-06-04; First posted 2021-06-23 (Actual); Last update posted 2022-03-24 (Actual); Status verified 2021-06

CONDITIONS: Neurodevelopmental Disorders; Emotional Disorder; Behavior Disorders
Keywords: Social and emotional learning; Social return on investment; Gamification; Behavioral and Emotional Disorders
MeSH Terms: conditions — Neurodevelopmental Disorders; Mental Disorders; Behavior | interventions — Methods

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Renew Intervention Group (Experimental): Participants in the group will receive training to help children strengthen social, emotional and behavioral knowledge and resilience.
  Interventions: Other: The RENEW Intervention
- Parallel Control Group (No Intervention): Participants in the group will receive the usual bible lessons and activities

INTERVENTIONS:
Other: The RENEW Intervention — An game-based intervention that will provide lessons and activities in social-awareness, self-management, self-awareness, relationships and decision making in effort to strengthen social, emotional and behavioral competence. The intervention will be administered tri-weekly for 20 minutes each session.
  Other Names: The Resilience in Emotional and Behavioral Wellbeing (RENEW) Intervention
  Arms: Renew Intervention Group

SUMMARY:
Behavioral and emotional disorders adversely affect overall health and well-being. Prevalence rates among children and adolescents classified with behavioral and emotional disorders or neurodevelopmental disorders (NDD), as recently redefined in ICD-11, have steadily increased over the past decade. In particular, prevalence rates among persons classified with Autism Spectrum Disorders (ASD), the fastest rising behavioral and emotional disorder, have sharply risen over the past five years and is now estimated at 1 in 54. Shared symptoms within behavioral and emotional disorders include persistent social, emotional and behavioral functioning deficits that often impact self-management, social-awareness and metacognition competences, in addition to adulthood health and wellness life course transition management.

Social and Emotional Learning (SEL) stakeholder advocates have contributed meaningfully to the strengthening of behavioral and emotional health through interventions that focus primarily on physical and mental health outcomes of diagnosed individuals. However, focus on spiritual health outcomes and the at-risk population remain largely underutilized. Research that seeks to employ an integrative physical-mental-spiritual approach to strengthen social, emotional and behavioral resilience, of at-risk school age populations where social stigma and prohibitive treatment costs remain barriers to treatment is needed to help expand the field's understanding of the reciprocal relationship between spiritual health and emotional and behavioral outcomes.

The RENEW (Resilience in Emotional and Behavioral Wellbeing) intervention will employ a multidisciplinary approach of social and emotional learning competency training, gamification principles and faith-centered values to strengthen social, behavioral and emotional resilience and competencies of those at risk for behavioral and emotional disorders, via a child-as co-researcher approach.

DETAILED DESCRIPTION:
Emotional and Behavior Disorders (EBD) or neurodevelopmental disorders (NDD) as recently redefined are a collection of behavioral and cognitive disorder classifications that describe a spectrum of deficits in social functioning, metacognition and self-management competencies, in particular, among children and adolescence. The subcategories of NDDs as listed in World Health Organization's 11th edition of the International Statistical Classification of Diseases and Related Health Problems (ICD) include Autism Spectrum Disorder (ASD), Attention-Deficit Hyperactivity Disorder (ADHD), Development of Learning Disorder and Disorders of Intellectual Development.

Prevalence rates among children and adolescents classified with EBDs or NDDs have steadily increased over the past decade. Autism Spectrum Disorders (ASD) or Autism Spectrum Conditions (ASC) is the fastest growing NDD affecting approximately one percent (1%) of the world's population. Prevalence rates among persons diagnosed with Autism Spectrum Conditions (ASC) have steadily risen over the past decade and are now estimated at 1 in 54. Autism's spectrum of social, emotional and behavioral impairments often range in severity and impact poor adulthood outcomes, primarily in health and wellness life course trajectories, of the unclassified. Shared symptoms within EBDs/NDDs include persistent social and behavioral functioning deficits that often impact self-management, social-awareness and metacognition competences, in addition to adulthood health and wellness life course transition management.

According to the World Health Organization (WHO), there are three main ways to classify health interventions, namely by target (the entity on which the action is carried out), action (a deed done by an actor to a target), or means (the process and methods by which the action is carried out). Empirical research has identified currently available social and emotional learning (SEL) interventions that target the clinically diagnosed. However, an issue with such interventions is that they provide no support to at-risk and/or undiagnosed behavioral and emotional disorder (EBD) vulnerable populations. The SEL intervention literature has also documented available psychosocial actions to support EBD children and young persons, such as cognitive behavioral therapy (CBT) and executive functioning skills training. However, a vulnerability of these actions is that they are often secular or void of a spiritual, religious or personal belief dimension to effect meaningful transformation as well as not participatory of EBD youth in the research process. Lastly, the SEL intervention literature has illuminated evidence on the available means/methods to support or deliver actions to EBD youth, such as via commercial-off-the-shelf (COTS) software, virtual reality (VR) technologies, games and robot-based platforms. However, a drawback of such means or methods is that they are often cost prohibitive, not conducive to facilitating citizen development and lacking in gamification features to strengthen end user engagement. Thus, there is a need to supplement the existing SEL intervention literature with programs that support spiritual health outcomes of at-risk EBD youth in a manner that fosters co-researcher opportunities and generates a social return on investment.

In this paper, we describe a protocol for a pilot evaluation of a faith-centered, non-medical, gamification assisted intervention, dubbed RENEW (Resilience in Emotional and Behavioral Wellbeing), an innovative, culturally appropriate, cost effective and participatory program developed to identify and strengthen social emotional behavioral resilience among primary and middle age school children populations who are increasingly exhibiting social emotional behavior symptoms. The research is situated at the intersection of technology, spirituality and global health practice in effort to strengthen contributions to health and wellness outputs, outcomes and impacts. The research endeavor will employ a multidisciplinary blend of gamification principles, co-researcher participation and faith-centered values to strengthen social, behavioral and emotional resilience competencies in effort to enhance social and behavioral deficit management.

ELIGIBILITY:
Inclusion Criteria:

* Home Internet access

Exclusion Criteria:

* No parental consent
* Sensory challenges to electronic devices

Ages: 8 Years to 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 60 (Estimated)
Dates: Start 2021-09-07 (Actual); Primary Completion 2022-03-30 (Estimated); Study Completion 2022-03-30 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in social-emotional competence on the Devereux Student Strengths Assessment - Mini instrument | Baseline and Week 10
  The Devereux Student Strengths Assessment - Mini is a 8-point brief version of the Devereux Student Strengths Assessment intended to serve as a universal screener of social and emotional competencies
  Rating Scale:
  (Never = 0; Rarely = 1; Occasionally = 2; Frequently = 3; Very Frequently = 4)
  High scores indicate a proficiency in social-emotional competence Low scores indicate need for instruction in social-emotional competence
Change from baseline in Self-Management assessment score on the Self-Management knowledge assessment form | Baseline and Week 6
  The Self-Management assessment is a 10-question quiz designed to assess a participants knowledge of self-management
  Rating Scale:
  (Need for knowledge of self-management < 60); (Average knowledge of self-management >= 60 and < 80); (Knowledge Proficiency of self-management >= 80)
  High scores indicate a proficiency in self-management knowledge Low scores indicate need for instruction in self-management knowledge
Change from baseline in Self-Awareness assessment score on the Self-Awareness knowledge assessment form | Baseline and Week 6
  The Self-Awareness assessment is a 10-question quiz designed to assess a participants knowledge of self-awareness
  Rating Scale:
  (Need for knowledge of self-awareness < 60); (Average knowledge of self-awareness >= 60 and < 80); (Knowledge Proficiency of self-awareness >= 80)
  High scores indicate a proficiency in self-awareness knowledge Low scores indicate need for instruction in self-awareness knowledge
Change from baseline in Social-Awareness assessment score on the social-awareness knowledge assessment form | Baseline and Week 8
  The Social-Awareness assessment is a 10-question quiz designed to assess a participants knowledge of social-awareness
  Rating Scale:
  (Need for knowledge of social-awareness < 60); (Average knowledge of social-awareness >= 60 and < 80); (Knowledge Proficiency of social-awareness >= 80)
  High scores indicate a proficiency in social-awareness knowledge Low scores indicate need for instruction in social-awareness knowledge
Change from baseline in Relationships assessment score on the relationships knowledge assessment form | Baseline and Week 8
  The Relationships assessment is a 10-question quiz designed to assess a participants knowledge of relationships
  Rating Scale:
  (Need for knowledge of relationships < 60); (Average knowledge of relationships >= 60 and < 80); (Knowledge Proficiency of relationships >= 80)
  High scores indicate a proficiency in relationship knowledge Low scores indicate need for instruction in relationship knowledge
Change from baseline in Decision-Making assessment score on the decision-making assessment form | Baseline and Week 10
  The Decision-Making assessment is a 10-question quiz designed to assess a participants knowledge of decision-making
  Rating Scale:
  (Need for knowledge of decision-making < 60); (Average knowledge of decision-making >= 60 and < 80); (Knowledge Proficiency of decision-making >= 80)
  High scores indicate a proficiency in decision-making knowledge Low scores indicate need for instruction in decision-making knowledge

SECONDARY OUTCOMES:
Change from baseline in Global self-concept score on the Social Emotional Assets and Resilience Scale - Child Short Form | Baseline to Week 10
  The Social Emotional Assets and Resilience Scale - Child Short form is a 12-question, self-report measure of a child's perception of his or her own global self-concept score.
  Rating Scale:
  (Never = 1; Sometimes = 2; Often = 3; Always = 4)
  High scores indicate adequacy in self-concept perception Low scores indicate inadequacy in self-concept perception

CONTACTS AND LOCATIONS:
Overall Officials: Usman Iqbal, PhD, Principal Investigator — Taipei Medical University
Locations (1):
- Taipei Adventist American School, Taipei, Shilin, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Garwood, J. D., Peltier, C., Sinclair, T., Eisel, H., McKenna, J. W., & Vannest, K. J. (2020). A Quantitative Synthesis of Intervention Research Published in Flagship EBD Journals: 2010 to 2019. Behavioral Disorders. https://doi.org/10.1177/0198742920961341
- [Result] Bitta M, Kariuki SM, Abubakar A, Newton CRJC. Burden of neurodevelopmental disorders in low and middle-income countries: A systematic review and meta-analysis. Wellcome Open Res. 2017 Dec 29;2:121. doi: 10.12688/wellcomeopenres.13540.3. eCollection 2017. PMID 29881784
- [Result] Fortune N, Madden R, Riley T, Short S. The International Classification of Health Interventions: an 'epistemic hub' for use in public health. Health Promot Int. 2021 Dec 23;36(6):1753-1764. doi: 10.1093/heapro/daab011. PMID 33585880
- [Result] Ketcheson L, Hauck JL, Ulrich D. The levels of physical activity and motor skills in young children with and without autism spectrum disorder, aged 2-5 years. Autism. 2018 May;22(4):414-423. doi: 10.1177/1362361316683889. Epub 2017 Mar 1. PMID 29152992
- [Result] Maenner MJ, Shaw KA, Baio J; EdS1; Washington A, Patrick M, DiRienzo M, Christensen DL, Wiggins LD, Pettygrove S, Andrews JG, Lopez M, Hudson A, Baroud T, Schwenk Y, White T, Rosenberg CR, Lee LC, Harrington RA, Huston M, Hewitt A; PhD-7; Esler A, Hall-Lande J, Poynter JN, Hallas-Muchow L, Constantino JN, Fitzgerald RT, Zahorodny W, Shenouda J, Daniels JL, Warren Z, Vehorn A, Salinas A, Durkin MS, Dietz PM. Prevalence of Autism Spectrum Disorder Among Children Aged 8 Years - Autism and Developmental Disabilities Monitoring Network, 11 Sites, United States, 2016. MMWR Surveill Summ. 2020 Mar 27;69(4):1-12. doi: 10.15585/mmwr.ss6904a1. PMID 32214087
- [Result] Price S. Addressing Autism: Giving Physicians Tools. Tex Med. 2019 Dec 1;115(12):42-44. PMID 31800089
- [Result] Wiggins LD, Durkin M, Esler A, Lee LC, Zahorodny W, Rice C, Yeargin-Allsopp M, Dowling NF, Hall-Lande J, Morrier MJ, Christensen D, Shenouda J, Baio J. Disparities in Documented Diagnoses of Autism Spectrum Disorder Based on Demographic, Individual, and Service Factors. Autism Res. 2020 Mar;13(3):464-473. doi: 10.1002/aur.2255. Epub 2019 Dec 23. PMID 31868321
- [Derived] Bowrin P, Bowrin E, Iqbal U, Sanna M. Benefits of RENEW: A Faith-Infused, Game-Based Social-Emotional Intervention: Evidence from a Pilot Cluster Randomized Crossover Trial on Primary School Children in Taiwan. J Relig Health. 2025 Jun;64(3):1594-1606. doi: 10.1007/s10943-024-02224-z. Epub 2024 Dec 24. PMID 39719545